CLINICAL TRIAL: NCT03341039
Title: PHIL Evaluation in the Endovascular Treatment of Intracranial Cerebral ArterioVenous Malformation a European Multi-center, Observational, Prospective, Single Arm and Open Label Study
Brief Title: PHIL Evaluation in the Endovascular Treatment of Intracranial Cerebral ArterioVenous Malformation (cAVM)
Status: Terminated | Type: Observational
Why Stopped: Termination of the study due to low enrolment
Sponsor: Microvention-Terumo, Inc. (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: cAVM-PHIL Registry
Record Dates: First submitted 2017-10-18; First posted 2017-11-14 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Cerebral AV Malformation
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of PHIL® liquid embolic agent in endovascular embolization of cerebral arteriovenous malformations.

DETAILED DESCRIPTION:
This is an European multi-center observational study. Treatments and follow-up visits will be done as per standard of care.

The objective of this study is to evaluate the efficacy and safety of the PHIL® device in the treatment of intracranial cerebral arteriovenous malformation. The PHIL® device, a non-adhesive liquid embolic agent, has been CE marked since July 2014. It is intended for use in the embolization of lesions in the peripheral and neurovasculature, including arteriovenous malformations and hypervascular tumors.

All patients with a cAVM, ruptured or unruptured, eligible for endovascular treatment with a liquid embolic agent, PHIL®, based on multidisciplinary consensus are eligible for this study. A maximum of 108 patients will be enrolled in 18 European Institutions.

The expected approximate study duration is 39 months.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a ruptured or unruptured and previously endovascularly untreated cAVM that are eligible for endovascular treatment with PHIL® alone or in conjunction with N-Butyl cyanoacrylate glue (NBCA) and/or coils (e.g. if "pressure cooking" technique is needed or used).
2. All patients with a previously endovascularly treated cAVM in which NBCA and/or coils (but not another non-adhesive liquid embolic agent) have been used may be included.**
3. All patients with a remaining cAVM, ruptured or unruptured, that has previously been treated with NS and/or RT may be included.
4. Patient or patient's legally authorized representative has received information about data collection and has signed and dated an Informed Consent Form. (Based on the country's regulation).

Exclusion Criteria:

1. cAVM not eligible for endovascular treatment
2. cAVM previously treated with a non-adhesive liquid embolic agent other than PHIL®
3. Treatment requiring the use of any other non-adhesive embolic liquid
4. Patient is allergic to iodine
5. Premature and newborn infant
6. Patient with renal failure or significant liver impairment
7. Patient is participating in another study evaluating other medical devices, other procedures or medications.
8. Any other condition that might prevent patient participation in the study or follow up
9. Patient does not want to and/or refuses to give consent to the collection and processing of data required for centralized monitoring

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a cAVM, ruptured or unruptured, eligible for endovascular treatment with a liquid embolic agent, PHIL®, based on multidisciplinary consensus.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Overall cure rate | immediately after final embolization
Cure rate with regard to the aim of the endovascular treatment | immediately after final embolization
Overall cure rate | 3-6 months
Cure rate with regard to the aim of the endovascular treatment | 3-6 months
Clinical outcome compared to baseline | up to 3 days
  Assessment by mRS
Clinical outcome compared to baseline | 1 month after each embolization
  Assessment by mRS
Clinical outcome compared to baseline | 3-6 months after the final embolization
  Assessment by mRS

SECONDARY OUTCOMES:
Adverse Events | 1 months after last embolization
  AE related to the PHIL procedure and/or to the techniques used during each embolization
Total volume of injected PHIL | during each embolization
Volume/superselective injection | during each embolization
Length of reflux of PHIL | during each embolization
Amount of pedicles catheterized | during each embolization
Overall injection time | during each embolization
Overall radiation dose given to the patient during EVT | during each embolization

CONTACTS AND LOCATIONS:
Locations (16):
- Rigshospitalet University, Copenhagen, Denmark
- France (5):
  - CHU Pellgrin, Bordeaux
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - La Fondation Rothschild, Paris
  - Hôpital Pierre Paul Riquet, Toulouse
- Spain (5):
  - Hospital Universitario General de Catalunya, Barcelona
  - Hospital Nuestra Senora del Rosario, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Universitetssjukhus Umea, Umeå
  - Uppsala University, Uppsala
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham
  - Western General Hospital, Edinburgh
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No